CLINICAL TRIAL: NCT02006563
Title: Evaluation of Metabolic Tumor Volumes in Radiation of Primary Brain Tumors
Brief Title: Metabolic Tumor Volumes in Radiation Treatment of Primary Brain Tumors
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Radka S. Stoyanova, Research Associate Professor, University of Miami
Other Study IDs: 20100809
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Brain Tumor; Glioblastoma Multiforme
Keywords: Brain Tumor; Glioblastoma multiforme; GBM; Metabolic Tumor Volume; MTV; Clinical Tumor Volume; CTV
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* Metabolic Tumor Volume (MTV), identified by Magnetic Resonance Spectroscopic Imaging (MRSI) is different from the Clinical Target Volume (CTV) used for radiation dose delivery in the treatment of brain tumors.
* If MTV > CTV, the investigators hypothesize that the difference in volumes (cc) is related to worse clinical outcome. Furthermore, in case of local recurrence, the lesion is located in the MTV area that is outside of the CTV.
* Alternatively, if CTV > MTV, then the difference in volumes is related to higher treatment toxicity.

DETAILED DESCRIPTION:
Metabolic Tumor Volume (MTV), identified by Magnetic Resonance Spectroscopic Imaging (MRSI) is different from the Clinical Target Volume (CTV) used for radiation dose delivery in the treatment of brain tumors.

* If MTV > CTV, the investigators hypothesize that the difference in volumes (cc) is related to worse clinical outcome. Furthermore, in case of local recurrence, the lesion is located in the MTV area that is outside of the CTV.
* Alternatively, if CTV > MTV, then the difference in volumes is related to higher treatment toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed primary brain tumor.
* Patients may be enrolled prior to surgery, after surgical resection or with unresectable tumors.
* Patients must be 18 years or older.
* Patients who do not have metal in the body (e.g. pacemakers, implants) that would preclude them from undergoing MRI/MRS exam
* Patients who do not suffer from claustrophobia (fear of enclosed spaces)
* Karnofsky performance status ≥ 60.
* Patients whose size would allow them to fit into the bore of the MRI instrument.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients younger than 18 years.
* Inability to undergo MRI/MRS exam because of metal in the head or body, such as implants, pacemaker, or biostimulation device. Claustrophobia (fear of enclosed spaces).
* Karnofsky performance status < 60.
* Patients too large (> 300 lbs.) to fit into the bore of the MRI instrument.
* Inability to understand the informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is estimated that approximately 39% of the patients with primary brain tumors, seen in the Department of Radiation Oncology, Sylvester Cancer Center are women. Further, it is estimated that 58% of patients are White, 6% are African American, 36% are Hispanic and 0% are other based upon standard NIH definitions.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2011-06-08 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Difference between Metabolic Tumor Volumes and Clinical Tumor Volumes in Patients with Brain Tumors | 2 years
  To evaluate the extent to which tumor volumes, determined by spectroscopic imaging (MTV) differ from the traditionally prescribed clinical treatment volumes (CTV) for radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Radka Stoyanova, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No